CLINICAL TRIAL: NCT03642665
Title: Frozen-thawed Embryo Transfer in a Natural Versus Artificial Cycle: a Randomized Clinical Trial
Brief Title: Natural Versus Artificial Cycle for Frozen-Thawed Embryo Transfer
Acronym: NAFT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: GZA Ziekenhuizen Campus Sint-Augustinus (Other); Imelda Hospital, Bonheiden (Other); Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S61372
Record Dates: First submitted 2018-07-17; First posted 2018-08-22 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-02

CONDITIONS: Embryo Transfer
MeSH Terms: interventions — Estradiol; Progesterone

STUDY DESIGN:
Intervention Model Description: Multicenter prospective randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Natural cycle (Experimental): no medication
  Interventions: Drug: Natural cycle
- Artificial cycle (Active Comparator): Oestradiol valerate (Progynova, Bayer, Germany) 6mg daily will be given from day 2 of the cycle. The dose of Progynova is increased to 8mg daily if the endometrial thickness is less than 7mm after 7-10 days of Progynova use. Progynova will be discontinued the day of the pregnancy test in case of a negative result. In case of a pregnancy, Progynova will be continued until 12 weeks or until diagnosis of a non-viable pregnancy.
  Micronized progesterone (Utrogestan, Besins, Belgium) 200 mg vaginally three times daily is started as soon as the endometrial thickness is 7 mm. Utrogestan will be discontinued the day of the pregnancy test in case of a negative result. In case of a pregnancy, Utrogestan will be continued until 12 weeks or until diagnosis of a non-viable pregnancy.
  Interventions: Drug: Estradiol Valerate; Drug: Micronized progesterone

INTERVENTIONS:
Drug: Natural cycle — no medication
  Arms: Natural cycle
Drug: Estradiol Valerate — Oestradiol valerate (Progynova, Bayer, Germany) 6mg daily will be given from day 2 of the cycle. The dose of Progynova is increased to 8mg daily if the endometrial thickness is less than 7mm after 7-10 days of Progynova use. Progynova will be discontinued the day of the pregnancy test in case of a negative result. In case of a pregnancy, Progynova will be continued until 12 weeks or until diagnosis of a non-viable pregnancy.
  Other Names: Artificial cycle
  Arms: Artificial cycle
Drug: Micronized progesterone — Micronized progesterone (Utrogestan, Besins, Belgium) 200 mg vaginally three times daily is started as soon as the endometrial thickness is 7 mm. Utrogestan will be discontinued the day of the pregnancy test in case of a negative result. In case of a pregnancy, Utrogestan will be continued until 12 weeks or until diagnosis of a non-viable pregnancy.
  Other Names: Artificial cycle
  Arms: Artificial cycle

SUMMARY:
This study evaluates clinical pregnancy rates, obstetrical outcome parameters, costs and patient preferences in natural cycle versus artificial cycle frozen embryo transfers (FET).

DETAILED DESCRIPTION:
Transfer of cryopreserved embryos can be performed in a natural cycle (NC-FET) or in an artificially prepared cycle (AC-FET). Both cycle regimens have their advantages and disadvantages. So far, most comparative studies have failed to identify the optimal protocol for FET. In this study patients undergoing FET will be randomized between an endometrial preparation by a natural cycle or by an artificial cycle (by oestradiol validate and micronized progesterone).

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing FET after a first, second or third fresh IVF/ICSI cycle
* Single embryo transfer (SET) or Double embryo transfer (DET)
* Female age between 18-45 year
* Women having a natural ovulatory cycle (24-35 days)
* Normal uterine cavity (fundal indentation at the cavity <10mm)
* Written informed consent

Exclusion Criteria:

* Use of donor gametes
* BMI > or equal to 35 kg / m2
* Any contra-indication to estrogen or progesterone supplementation (e.g. history of thrombosis, prior or current hormone-sensitive malignancy…)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 554 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate with fetal heart beat | 9 weeks
  Clinical pregnancy rate with fetal heart beat diagnosed by ultrasound no later than the gestational age of 9 weeks

SECONDARY OUTCOMES:
Biochemical pregnancy rate | 9 weeks
Miscarriage rate | 12 weeks
Ectopic pregnancy rate | 9 weeks
Live birth rate | 41 weeks
Multiple pregnancy rate | 9 weeks
Adverse events | 12 weeks
  tombo-embolic events, serious side-effects (car leaflet) which require cancellation of treatment
Cycle cancellation rate | 4 weeks
Endometrial thickness | 3 weeks
Endometrial pattern | 3 weeks
  Sonographic aspect of the endometrium (triple-line, no triple-line)
number of center visits to monitor FET cycle | From date of randomization until the date of the embryo transfer or until cancellation (estimated period of time up to 4 weeks)
cost analysis per treatment cycle | From date of randomization until the date of the embryo transfer or until cancellation (estimated period of time up to 4 weeks)
patient satisfaction | 12 weeks
  To evaluate the effect of the different regimens on patients wellbeing/distress, Patient Reported Experience Measures (PREMS) from validated questionnaires will be used. Twenty-two questions from the Benyamini questionnaire will be used (Benyamini et al. 2005) and 10 questions from the subscales 'environment' (α=0.81) and 'tolerability' (α=0.75) of the FertilQol questionnaire (Pedro et al 2013). On the day of embryo transfer, the treating gynecologist will hand out the questionnaire to the patient. The patient will return the filled-in questionnaire on the day of the pregnancy test, before she knows the result of the pregnancy test.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No